CLINICAL TRIAL: NCT05342220
Title: Effect of Ischemic Preconditioning on Relapse of Nonvalvular Atrial Fibrillation After Electrocardioversion
Brief Title: Effect of Ischemic Preconditioning on Atrial Fibrillation After Electrocardioversion
Acronym: PRECON-AF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Josefs-Hospital Wiesbaden GmbH (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PRECON
Record Dates: First submitted 2022-04-06; First posted 2022-04-22 (Actual); Last update posted 2024-07-09 (Actual); Status verified 2024-07

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Remote Ischemic Preconditioning (Active Comparator): Remote ischemic preconditioining
  Interventions: Procedure: Remote ischemic preconditioning
- Control (Sham Comparator): Sham preconditioning
  Interventions: Procedure: Sham preconditioning

INTERVENTIONS:
Procedure: Remote ischemic preconditioning — Remote ischemic preconditioning through inflation of a blood pressure cuff to pressure values > 200mmHg for 5 minutes followed by 5 minutes of reperfusion (3 times each) before electrocardioversion Electrical cardioversion for atrial fibrillation (100, 150, 200 Joule)
  Arms: Remote Ischemic Preconditioning
Procedure: Sham preconditioning — Inflation of a blood pressure cuff to pressure values ~ 10mmHg for 5 minutes followed by 5 minutes of reperfusion (3 times each) before electrocardioversion
  Arms: Control

SUMMARY:
Remote ischemic preconditioning is one way to influence the success of therapy in cardiovascular patients. By means of remote ischemic preconditioning the incidence of atrial fibrillation after cardiac surgery was reduced by 54%. The investigators aim to investigate the effect of ischemic preconditioning in an easy-to-perform protocol with regard to the recurrence of atrial fibrillation after electrical cardioversion.

ELIGIBILITY:
Inclusion Criteria:

* Patients with paroxysmal or persistent atrial fibrillation who give written informed consent to participate in the study
* Age > 18 years
* Consent capacity

Exclusion Criteria:

* Age under 18 years
* Pregnancy
* Lack of consent capacity

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2024-03-31 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Number of subjects with recurrence of atrial fibrillation 30 days after electrical cardioversion | 30 days

SECONDARY OUTCOMES:
Number of patients with short-term cardioversion success | 30 seconds
  Sinus rhythm lasting > 30 seconds after electrocardioversion
Minimum energy required for successful electrocardioversion (in Joule) | 30 days
Cumulative energy applied for successfull electrocardioversion (in Joule) | 30 days
Cumulative number of shocks delivered for successfull electrocardioversion | 30 days
Number of patients experiencing death from any cause, stroke /transient ischemic attack, relevant post-ECV arrhythmia and procedure-associated complications | 30 days
  Safety endpoint

CONTACTS AND LOCATIONS:
Locations (1):
- St. Josefs-Hospital Wiesbaden, Wiesbaden, Hesse, Germany

REFERENCES:
- [Derived] Keim C, Wiedenmann L, Schubert T, Rothe M, Dobre BC, Kaess BM, Ehrlich JR, Boehmer AA. Remote Ischemic Preconditioning for Electrical Cardioversion of Atrial Fibrillation-the Prospective Randomized PRECON-AF Study. CJC Open. 2025 Mar 10;7(5):571-578. doi: 10.1016/j.cjco.2025.03.004. eCollection 2025 May. PMID 40433224